CLINICAL TRIAL: NCT03529981
Title: Wearable Emotion Prosthetics for Post Traumatic Stress Disorder
Acronym: EP-PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Greg Siegle, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: PRO17110107
Record Dates: First submitted 2018-04-16; First posted 2018-05-21 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Health Behavior
Keywords: PTSD
MeSH Terms: conditions — Health Behavior; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: randomized, controlled factorial within subject design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: On-demand intervention was provided on only some physiologically detected stress events
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stress incidents without TVS (Active Comparator): a fraction of physiological detected stress incidents will not trigger TVS
  Interventions: Other: no active intervention
- TVS in response to participant initiation or stress detection (Experimental): The majority of detected stress incidents will trigger TVS. Participants can also trigger TVS voluntarily
  Interventions: Other: Tuned Vibroacoustic Stimulation (TVS)

INTERVENTIONS:
Other: Tuned Vibroacoustic Stimulation (TVS) — TVS is an exteroceptive cue that may reduce subjective and physiological indicators of stress and increase behavioral performance
  Arms: TVS in response to participant initiation or stress detection
Other: no active intervention — No intervention will be administered
  Arms: Stress incidents without TVS

SUMMARY:
Involuntary stress reactions including hyper-reactivity and dissociation are key diagnostic features of many psychiatric disorders, are difficult to treat, and predict poor outcomes in conventional and neurobehavioral interventions. Here, we evaluate the extent to which a novel intervention, Tuned Vibroacoustic Stimulation (TVS), capitalizing on a preserved neurocircuitry for sympathetic and parasympathetic system activity can be used to modify arousal responses, overriding otherwise prepotent negative stress reactions.

PTSD has been characterized by dysregulated responses to stress as a result of severe acute or chronic trauma resulting in significantly impaired functioning, quality of life, and morbidity/mortality. Physiologically, PTSD severity has been associated with elevated sympathetic tone and low heart rate variability suggesting that parasympathetic tone is suppressed. Lower heart rate variability specifically, as a measure of parasympathetic tone, is closely associated with impaired performance and resilience. In our first study (in review), we showed that in some individuals, TVS is associated with increased heart rate variability and performance under stress along with reduced subjective stress. These results suggest that TVS could provide some therapeutic benefit in PTSD.

N=100 individuals with mild-moderate PTSD (as assessed by PCL-5/CAP5), at least half of which are military Veterans, will be assessed physiologically during active interventions. Mechanisms of attentional focus on cognitive and emotional stimuli will be assessed. Participants will also have a real-world intervention to determine if TVS helps alleviate stress, symptoms, and medication burden in the real world when stress has been identified. Success will suggest a new intervention pathway for a traditionally treatment-resistant dimension of psychopathology.

DETAILED DESCRIPTION:
This protocol will examine and elucidate a mechanistic model for tuned vibroacoustic stimulation (TVS), an exteroceptive cue that has been shown to reduce subjective and physiological indicators of stress and increase behavioral performance in healthy subjects. In this study, we will test whether TVS can reduce subjective and physiological signs of stress, improve performance, alleviate symptoms, and reduce medication burden in adults with post-traumatic stress disorder (PTSD). This protocol will also examine whether software that cues TVS in response to biological stress markers helps users detect, regulate, and develop long-term resilience to stress outside of the laboratory.

Aim 1: Examine how TVS alters calmness and stress markers. Our overall hypothesis is that TVS, in combination with some other task, increases performance on that task by decreasing stress and increasing emotion regulation.

Hypothesis 1: TVS during an attention task will lead to decreased GSR, increased HRV, and increases in prefrontal gamma and theta band EEG, along with improved behavioral performance on a focused attention, working memory and emotional information processing task. TVS will also reduce subjective stress levels.

Aim 2: Examine the extent to which software, which monitors real time biological stress markers of users, and in response, automatically signals wearable hardware to deliver TVS when user is stressed, will be able to help users detect, regulate, and develop long-term resilience to stress outside the laboratory for two weeks.

Hypothesis 2.1: Evaluate whether subjects with PTSD in the real world will use our software to detect and alert them of stress dynamically and if this is associated with stress regulation.

Hypothesis 2.2: Examine whether TVS is associated with stress regulation. Hypothesis 2.3: Examine whether TVS is associated with reduction in PTSD symptoms and, possibly, medication burden.

Over 39 million Americans suffer from excessive chronic stress, which can be psychologically and physically debilitating (Salleh, 2008). Untreated chronic stress plays a role in the development of major illnesses such as cardiovascular disease, obesity, anxiety and depression (Dallman et al., 2006; Swaab, Bao, & Lucassen, 2005). Post-traumatic stress disorder (PTSD), is a severe mental illness that impacts millions of veterans and civilians nationwide. Existing treatments for chronic stress and PTSD are often ineffective, have adverse effects, and are prohibited by cost, time-commitment, and accessibility, resulting in high rates of substance abuse and suicide (Jonas et al., 2013; Watts et al., 2013). Stress in general, and PTSD more specifically, are characterized by hyper-reactivity in the sympathetic nervous system which is associated with increased arousal and vigilance, and compromised reactivity of the parasympathetic nervous system, which helps to regulate emotion and stress responses (Kibler, Tursich, Ma, Malcolm, & Greenbarg, 2014; Lehrer & Gevirtz, 2014).

PTSD has been characterized by dysregulated responses to stress as a result of severe acute or chronic trauma resulting in significantly impaired functioning, quality of life, and morbidity/mortality. Physiologically, PTSD severity has been associated with elevated sympathetic tone and low heart rate variability suggesting that parasympathetic tone is suppressed. HRV is widely used as a biomarker for the coordinated activity of the sympathetic and parasympathetic nervous symptom. A calmer, less stressful state is typically marked by increased HRV, likely attributed to respiration based parasympathetic stimulation (Grossman & Taylor, 2007). GSR is also a reliable index for sweat gland activity and changes in activation level of the sympathetic nervous system, and GSR usually increases with higher levels of stress (Mohan, Sharma, & Bijlani, 2011). EEG changes, such as elevated prefrontal gamma and theta, have also been associated with state of relaxed alertness. Our initial data (submitted) suggest that for some individuals, TVS can boost heart rate variability and performance under stress while reducing subjective stress. These results suggest that TVS could provide some therapeutic benefit in PTSD.

Large scientific literature supports the role of vibration in regulating stress physiology (Takahashi, Ohashi, & Yokoyama, 2011; M. Uchikune, 2002; M. Uchikune, 2004). For example, slow whole-body vibration, in the 0.01 to 0.3 Hz range, is associated with increased ratings of pleasantness and increased parasympathetic tone (M. Uchikune, 2002; M. Uchikune, 2004). Stimulation at about 100 Hz has been shown to activate the posterior insula (Coghill et al., 1994) which is associated with increased attention to interoception, as promoted in many meditative traditions. Transcutaneous targets for the vibration frequencies have also been identified, including stellate ganglion and vagus nerve (Cipriano et al., 2014; Fang et al., 2016).

In this study, we will be testing the potential for TVS to increase well-being (subjective calmness, increased performance, and physiological reactivity) in the PTSD population. Positive results would suggest that reduction in symptomatology may be possible without effort, and in lieu of specific interventions with medications or psychotherapy. A wearable form of TVS technology will be examined in a real-world setting. We will use ambulatory assessment to detect physiological indications of stress unique to each user and to provide user-optimized TVS, examining whether it increases parasympathetic nervous system reactivity in response to stress, thus decreasing subjective stress just as a user's stress begins to increase.

ELIGIBILITY:
Inclusion Criteria:

* Male/female who are 18 - 58 years of age
* For PTSD participants, must meet current DSM-V criteria for PTSD based on the PCL-5 (Score > 33) and MINI PTSD Scale (administered in lab).
* If taking psychoactive medications, must be on a stable regimen for 3 weeks or more.
* Must have a functioning smartphone with Apple iOS or Android

Exclusion Criteria:

* Refusal or inability to provide informed consent
* Current suicidal or homicidal ideation with intent and/or plan that, in the judgment of the investigator, should be the focus of treatment.
* Current or recent (within the last 8 weeks) physically aggressive behavior.
* Meets current DSM-V criteria for substance dependence ((serious substance use in DSM-V parlance, not in remission) except nicotine and caffeine), traumatic brain injury, bipolar affective disorder, schizophrenia or any psychotic disorder.
* Has unstable or serious medical illness, including history of stroke, epileptic disorder, or unstable cardiac disease, that would interfere with participation in treatment.
* Taking medications that could affect thinking which must be taken on the day of testing, or dependence on psychoactive drugs (prescription or non-prescription) that could affect thinking. That is, participants need to be able to think clearly to complete the proposed information processing tasks. And they need to be able to learn to be able to make use of the intervention. Examples of drugs which could affect performance on cognitive tasks or the administered physiological measures include beta-blockers, benzodiazepines, antipsychotics, stimulants (except for treatment of ADD/ADHD), narcotics, and anti--Parkinsonian drugs.
* Severe cognitive impairment or severe trauma
* Unable to comprehend or communicate in English, and unable to complete questionnaires written in English.
* Having any eye problems or difficulties in corrected vision or hearing, including poor color vision
* Having a North American Adult Reading Test (NAART) equivalent FSIQ < 85
* Severe or poorly controlled concurrent medical disorders or require medication that could cause negative thinking

Specific Exclusions for acoustic vibration include:

-- Any electrical implant (pacemaker, vagus nerve stimulator, etc).

Ages: 18 Years to 58 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2021-12-18 (Actual); Study Completion 2021-12-18 (Actual)

PRIMARY OUTCOMES:
Change in symptom ratings from pre- to post- | Change in symptom ratings over the approximately two weeks of the acute intervention (pre- to post- assessment)
  Subjective affect / symptom ratings will be obtained daily. Spline fitting will be used to create a smoothed estimate of trajectory, the beginning and end points of which will be compared.
Change in resting Heart Rate Variability (HRV) from pre- to post- | HRV will be measured during the entire study which is two weeks
  HRV, an index of parasympathetic reactivity, will be obtained throughout the day during the study. Increased HRV indicates increased parasympathetic reactivity, which suggests an increased physiological indicator of emotion regulation. Spline fitting will be used to create a smoothed estimate of trajectory, the beginning and end points of which will be compared.

SECONDARY OUTCOMES:
Change in Heart Rate Variability (HRV) during information processing tasks (composite) | HRV will be measured during the approximately 1 hour of information processing tasks, which will be administered approximately 2 weeks apart, at the pre- and post- intervention assessment visits.
  HRV, an index of parasympathetic reactivity, will be obtained during laboratory information processing tasks (paced auditory serial attention, emotional picture viewing). Increased HRV indicates increased parasympathetic reactivity, which suggests an increased physiological indicator of emotion regulation.
Galvanic skin response (GSR) during information processing tasks (composite) | GSR will be measured during the approximately 1 hour of information processing tasks, which will be administered approximately 2 weeks apart, at the pre- and post- intervention assessment visits.
  GSR, index of sympathetic reactivity, will be obtained during lab tasks before and after the intervention. Decreased GSR indicates decreased sympathetic reactivity, which suggests an increased physiological indicator of emotion regulation.
prefrontal gamma band EEG during information processing tasks (composite) | EEG will be measured during the approximately 1 hour of information processing tasks, which will be administered approximately 2 weeks apart, at the pre- and post- intervention assessment visits.
  prefrontal gamma band EEG will be obtained during lab information processing tasks. Increased prefrontal gamma band EEG suggests an increased physiological indicator of emotion regulation.

CONTACTS AND LOCATIONS:
Overall Officials: Greg Siegle, MD, Principal Investigator — Western Psychiatric Institute and Clinic
Locations (1):
- Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Following publication of primary results, individual anonymized data on primary outcome measures will be made available to other researchers. Before publication, primary outcome measures will be shared in negotiation with a proposed analysis plan from qualified investigators.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Following publication - available to all. Before publication - upon negotiation with qualified investigators
Access Criteria: Before publication - available in negotiation with Greg Siegle (gsiegle@pitt.edu). After publication the location of a data repository will be listed

REFERENCES:
- [Background] Brown KW, Ryan RM. The benefits of being present: mindfulness and its role in psychological well-being. J Pers Soc Psychol. 2003 Apr;84(4):822-48. doi: 10.1037/0022-3514.84.4.822. PMID 12703651
- [Background] Carlson LE, Brown KW. Validation of the Mindful Attention Awareness Scale in a cancer population. J Psychosom Res. 2005 Jan;58(1):29-33. doi: 10.1016/j.jpsychores.2004.04.366. PMID 15771867
- [Background] Cipriano G Jr, Neder JA, Umpierre D, Arena R, Vieira PJ, Chiappa AM, Ribeiro JP, Chiappa GR. Sympathetic ganglion transcutaneous electrical nerve stimulation after coronary artery bypass graft surgery improves femoral blood flow and exercise tolerance. J Appl Physiol (1985). 2014 Sep 15;117(6):633-8. doi: 10.1152/japplphysiol.00993.2013. Epub 2014 Aug 7. PMID 25103974
- [Background] Coghill RC, Talbot JD, Evans AC, Meyer E, Gjedde A, Bushnell MC, Duncan GH. Distributed processing of pain and vibration by the human brain. J Neurosci. 1994 Jul;14(7):4095-108. doi: 10.1523/JNEUROSCI.14-07-04095.1994. PMID 8027764
- [Background] Creswell JD. Mindfulness Interventions. Annu Rev Psychol. 2017 Jan 3;68:491-516. doi: 10.1146/annurev-psych-042716-051139. Epub 2016 Sep 28. PMID 27687118
- [Background] Dallman MF, Pecoraro NC, La Fleur SE, Warne JP, Ginsberg AB, Akana SF, Laugero KC, Houshyar H, Strack AM, Bhatnagar S, Bell ME. Glucocorticoids, chronic stress, and obesity. Prog Brain Res. 2006;153:75-105. doi: 10.1016/S0079-6123(06)53004-3. PMID 16876569
- [Background] Dittrich A. The standardized psychometric assessment of altered states of consciousness (ASCs) in humans. Pharmacopsychiatry. 1998 Jul;31 Suppl 2:80-4. doi: 10.1055/s-2007-979351. PMID 9754838
- [Background] Fang J, Rong P, Hong Y, Fan Y, Liu J, Wang H, Zhang G, Chen X, Shi S, Wang L, Liu R, Hwang J, Li Z, Tao J, Wang Y, Zhu B, Kong J. Transcutaneous Vagus Nerve Stimulation Modulates Default Mode Network in Major Depressive Disorder. Biol Psychiatry. 2016 Feb 15;79(4):266-73. doi: 10.1016/j.biopsych.2015.03.025. Epub 2015 Apr 2. PMID 25963932
- [Background] Fredrickson BL. The broaden-and-build theory of positive emotions. Philos Trans R Soc Lond B Biol Sci. 2004 Sep 29;359(1449):1367-78. doi: 10.1098/rstb.2004.1512. PMID 15347528
- [Background] Fredrickson BL, Branigan C. Positive emotions broaden the scope of attention and thought-action repertoires. Cogn Emot. 2005 May 1;19(3):313-332. doi: 10.1080/02699930441000238. PMID 21852891
- [Background] Fredrickson BL, Joiner T. Positive emotions trigger upward spirals toward emotional well-being. Psychol Sci. 2002 Mar;13(2):172-5. doi: 10.1111/1467-9280.00431. PMID 11934003
- [Background] Fredrickson BL, Levenson RW. Positive Emotions Speed Recovery from the Cardiovascular Sequelae of Negative Emotions. Cogn Emot. 1998 Mar 1;12(2):191-220. doi: 10.1080/026999398379718. PMID 21852890
- [Background] Fredrickson BL, Tugade MM, Waugh CE, Larkin GR. What good are positive emotions in crises? A prospective study of resilience and emotions following the terrorist attacks on the United States on September 11th, 2001. J Pers Soc Psychol. 2003 Feb;84(2):365-76. doi: 10.1037//0022-3514.84.2.365. PMID 12585810
- [Background] Grossman P, Taylor EW. Toward understanding respiratory sinus arrhythmia: relations to cardiac vagal tone, evolution and biobehavioral functions. Biol Psychol. 2007 Feb;74(2):263-85. doi: 10.1016/j.biopsycho.2005.11.014. Epub 2006 Nov 1. PMID 17081672
- [Background] Jonas DE, Cusack K, Forneris CA, Wilkins TM, Sonis J, Middleton JC, Feltner C, Meredith D, Cavanaugh J, Brownley KA, Olmsted KR, Greenblatt A, Weil A, Gaynes BN. Psychological and Pharmacological Treatments for Adults With Posttraumatic Stress Disorder (PTSD) [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2013 Apr. Report No.: 13-EHC011-EF. Available from http://www.ncbi.nlm.nih.gov/books/NBK137702/ PMID 23658937
- [Background] Kabat-Zinn J. An outpatient program in behavioral medicine for chronic pain patients based on the practice of mindfulness meditation: theoretical considerations and preliminary results. Gen Hosp Psychiatry. 1982 Apr;4(1):33-47. doi: 10.1016/0163-8343(82)90026-3. PMID 7042457
- [Background] Kabat-Zinn J, Massion AO, Kristeller J, Peterson LG, Fletcher KE, Pbert L, Lenderking WR, Santorelli SF. Effectiveness of a meditation-based stress reduction program in the treatment of anxiety disorders. Am J Psychiatry. 1992 Jul;149(7):936-43. doi: 10.1176/ajp.149.7.936. PMID 1609875
- [Background] Kibler JL, Tursich M, Ma M, Malcolm L, Greenbarg R. Metabolic, autonomic and immune markers for cardiovascular disease in posttraumatic stress disorder. World J Cardiol. 2014 Jun 26;6(6):455-61. doi: 10.4330/wjc.v6.i6.455. PMID 24976918
- [Background] Kok BE, Coffey KA, Cohn MA, Catalino LI, Vacharkulksemsuk T, Algoe SB, Brantley M, Fredrickson BL. How positive emotions build physical health: perceived positive social connections account for the upward spiral between positive emotions and vagal tone. Psychol Sci. 2013 Jul 1;24(7):1123-32. doi: 10.1177/0956797612470827. Epub 2013 May 6. PMID 23649562
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Lehrer PM, Gevirtz R. Heart rate variability biofeedback: how and why does it work? Front Psychol. 2014 Jul 21;5:756. doi: 10.3389/fpsyg.2014.00756. eCollection 2014. PMID 25101026
- [Background] Lomas T, Ivtzan I, Fu CH. A systematic review of the neurophysiology of mindfulness on EEG oscillations. Neurosci Biobehav Rev. 2015 Oct;57:401-10. doi: 10.1016/j.neubiorev.2015.09.018. Epub 2015 Oct 9. PMID 26441373
- [Background] Ludwig DS, Kabat-Zinn J. Mindfulness in medicine. JAMA. 2008 Sep 17;300(11):1350-2. doi: 10.1001/jama.300.11.1350. No abstract available. PMID 18799450
- [Background] Mohan A, Sharma R, Bijlani RL. Effect of meditation on stress-induced changes in cognitive functions. J Altern Complement Med. 2011 Mar;17(3):207-12. doi: 10.1089/acm.2010.0142. Epub 2011 Mar 9. PMID 21417807
- [Background] Ong AD, Bergeman CS, Bisconti TL, Wallace KA. Psychological resilience, positive emotions, and successful adaptation to stress in later life. J Pers Soc Psychol. 2006 Oct;91(4):730-49. doi: 10.1037/0022-3514.91.4.730. PMID 17014296
- [Background] Salleh MR. Life event, stress and illness. Malays J Med Sci. 2008 Oct;15(4):9-18. PMID 22589633
- [Background] Schofield TP, Creswell JD, Denson TF. Brief mindfulness induction reduces inattentional blindness. Conscious Cogn. 2015 Dec;37:63-70. doi: 10.1016/j.concog.2015.08.007. Epub 2015 Aug 28. PMID 26320867
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] Swaab DF, Bao AM, Lucassen PJ. The stress system in the human brain in depression and neurodegeneration. Ageing Res Rev. 2005 May;4(2):141-94. doi: 10.1016/j.arr.2005.03.003. PMID 15996533
- [Background] Takahashi I, Ohashi H, Yokoyama K. Optimum arousal level preservation system using biosignals. J Hum Ergol (Tokyo). 2011 Dec;40(1-2):119-28. PMID 25665216
- [Background] Teasdale JD, Segal ZV, Williams JM, Ridgeway VA, Soulsby JM, Lau MA. Prevention of relapse/recurrence in major depression by mindfulness-based cognitive therapy. J Consult Clin Psychol. 2000 Aug;68(4):615-23. doi: 10.1037//0022-006x.68.4.615. PMID 10965637
- [Background] Tugade MM, Fredrickson BL. Resilient individuals use positive emotions to bounce back from negative emotional experiences. J Pers Soc Psychol. 2004 Feb;86(2):320-33. doi: 10.1037/0022-3514.86.2.320. PMID 14769087
- [Background] Uttl B. North American Adult Reading Test: age norms, reliability, and validity. J Clin Exp Neuropsychol. 2002 Dec;24(8):1123-37. doi: 10.1076/jcen.24.8.1123.8375. PMID 12650237
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Watts BV, Schnurr PP, Mayo L, Young-Xu Y, Weeks WB, Friedman MJ. Meta-analysis of the efficacy of treatments for posttraumatic stress disorder. J Clin Psychiatry. 2013 Jun;74(6):e541-50. doi: 10.4088/JCP.12r08225. PMID 23842024
- [Background] Westbrook C, Creswell JD, Tabibnia G, Julson E, Kober H, Tindle HA. Mindful attention reduces neural and self-reported cue-induced craving in smokers. Soc Cogn Affect Neurosci. 2013 Jan;8(1):73-84. doi: 10.1093/scan/nsr076. Epub 2011 Nov 22. PMID 22114078
- [Result] Azam MA, Katz J, Mohabir V, Ritvo P. Individuals with tension and migraine headaches exhibit increased heart rate variability during post-stress mindfulness meditation practice but a decrease during a post-stress control condition - A randomized, controlled experiment. Int J Psychophysiol. 2016 Dec;110:66-74. doi: 10.1016/j.ijpsycho.2016.10.011. Epub 2016 Oct 18. PMID 27769879

DOCUMENTS (3):
  • Study Protocol (2018-05-07): https://cdn.clinicaltrials.gov/large-docs/81/NCT03529981/Prot_001.pdf
  • Statistical Analysis Plan (2018-05-07): https://cdn.clinicaltrials.gov/large-docs/81/NCT03529981/SAP_002.pdf
  • Informed Consent Form (2018-04-02): https://cdn.clinicaltrials.gov/large-docs/81/NCT03529981/ICF_000.pdf